CLINICAL TRIAL: NCT03069521
Title: Prospective, Feasibility Study to Evaluate the Safety of the EndoArt™ for Treatment of Subjects Suffering From Corneal Edema
Brief Title: Study to Evaluate the Safety of the EndoArt™ for Treatment of Subjects Suffering From Corneal Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye-yon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ECL00041
Record Dates: First submitted 2017-02-19; First posted 2017-03-03 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Chronic Cornel Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EndoArt® (Other): EndoArt® Artificial Endothelial Layer
  Interventions: Device: EndoArt® Artificial Endothelial Layer

INTERVENTIONS:
Device: EndoArt® Artificial Endothelial Layer — device is intended for use as an endothelial kearatoprosthesis

SUMMARY:
Prospective, feasibility study to evaluate the safety of the EndoArt® for treatment of 30 subjects suffering from corneal edema. Followed up for 12 months.

DETAILED DESCRIPTION:
Title: Prospective, feasibility study to evaluate the safety of the EndoArt® for treatment of subjects suffering from corneal edema

Device: EndoArt® (Artificial Endothelial Layer)

Intended Use: The EndoArt® device is intended for use as an endothelial kearatoprosthesis in patients with chronic cornel edema

Study Design: Prospective open-label feasibility clinical study

Study Objectives: To evaluate the safety of the EndoArt® implanted in subjects suffering from corneal edema.

Study Hypothesis: Treatment with the EndoArt® is safe and may result in alleviating symptoms resulting from chronic corneal edema (corneal thickness).

Study population: Men and women suffering from a decrease in vision due to chronic corneal edema that meet the inclusion/exclusion criteria and provide written Informed Consent will enrolled in the study.

Enrollment: A total of up to 30 subjects will be enrolled.

Study Duration: Completion of active enrollment is anticipated to last approximately 18 months. The primary end point will be achieved when the final study subject has completed 6 month follow up. Subject will be followed up to 12 month.

Primary Safety Endpoint: The frequency and severity of all treatment-related adverse events, during and after implantation of the EndoArt® and throughout the 6 month follow-up period. Adverse events will be assessed on a continuous basis from the procedure through the study completion at 6 months. Related adverse events include: corneal perforation, melting, uncontrolled inflammation, severe infection.

Secondary Efficacy Endpoints: Corneal thickness, Subjective corneal clarity, Pain as assessed by a Visual Analogue Scale (VAS) Measurement Best Corrected Distance Visual Acuity (BCDVA)

Study Treatment: Subjects will be implanted with the EndoArt®

ELIGIBILITY:
Inclusion Criteria:

1. Subject is over 40 years old
2. Subject with chronic corneal edema.
3. Subject with corneal thickness >650 µm
4. Subject with visual acuity 6/30 or worse (equivalent ETDRS)
5. Subject with better visual acuity in the contralateral eye.
6. Pseudophakic subject (anterior or posterior) with stable IOL.
7. Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed.

Exclusion Criteria:

1. Subject with best corrected visual acuity of 6/30 or worse in the fellow eye
2. Subject with history of ocular Herpes keratitis
3. Subject with severely scarred cornea (unfit for regular endothelial keratoplasty)
4. Subject with irregular posterior cornea (e.g. post PKP)
5. Subject who is suffering from infection of the cornea
6. Patients with band keratopathy and/or limbal stem cell deficiency.
7. Subject with clinical moderate to severe dry eye
8. Subject with phthisis or phthisis suspect
9. Subject with low ocular pressure ≤6 mmHg or higher than 25 mmHg.
10. Subject with aphakica
11. Subject with pseudophakodonesis
12. Subject with large iris defect which can compromise intraoperative AC stability.
13. Subjects after corneal refractive surgery.
14. Subject with glaucoma shunt (e.g. Ahmend valve)
15. Subject with neurotrophic corneal history
16. Subject with history of persistent corneal erosion difficulties with epithelial growth (re-epithelization)
17. Subject who is currently participating or have participated in an investigational study, other than this study, within the past 60 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Treatment-related adverse events | 6 months following EndoArt implantaion
  frequency and severity of all treatment-related adverse events

SECONDARY OUTCOMES:
Subjective corneal clarity | 12 months following EndoArt implantaion
  corneal clarity will be graded by the investigator.
  Scoring is as follow:
  * 0- clear
  * 1-iris details can be seen
  * 2- iris details are obscure
  * 3- can hardly see the pupil
  * 4- pupil or iris details ca not be seen
Pain as assessed by a Visual Analogue Scale (VAS) | 12 months following EndoArt implantaion
  VAS is a horizontal line, 100 mm in length, anchored by word descriptors at each end.
  The subject marks on the line the point that he feels represents his perception of his current state.
Measurement Best Corrected Distance Visual Acuity (BCDVA) | 12 months following EndoArt implantaion
  Visual acuity on the distance chart with best manifest correction for that distance
Corneal thickness | 12 months following EndoArt implantaion
  Corneal thickness will be measured by anterior segment Optical Coherence Tomography (OCT).

CONTACTS AND LOCATIONS:
Locations (8):
- International Vision Correction Research Centre (IVCRC) Universitätsklinikum Heidelberg, Heidelberg, Germany
- Israel (5):
  - Barzilai MC, Ashkelon
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Assuta Medical Center, Tel Aviv
  - Tel Aviv Souraski Medical Center, Tel Aviv
- AMC, Amsterdam, Netherlands
- IMO - Institut de Microcirurgia Ocular, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No